CLINICAL TRIAL: NCT01274741
Title: Pilot Study of an Integrated Exposure-Based Model for Posttraumatic Stress Disorder and Substance Use Disorder
Brief Title: Present- Versus Past-focused Therapy for PTSD and Substance Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Krinsley, PTSD Section Chief, VA Boston Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLA-CX000308-01 (VA CSRD)
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Posttraumatic Stress Disorder; Substance Use Disorder; Alcohol Use Disorder
Keywords: Posttraumatic stress disorder; Substance use disorder; Treatment efficacy; Randomized trial; Trauma; Substance abuse; Addiction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Alcoholism; Wounds and Injuries; Behavior, Addictive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seeking Safety (SS) (Active Comparator): 17 sessions of present-focused therapy Seeking Safety
  Interventions: Behavioral: Seeking Safety (SS)
- Creating Change (CC) (Experimental): 17 sessions of past-focused Creating Change
  Interventions: Behavioral: Creating Change (CC)

INTERVENTIONS:
Behavioral: Creating Change (CC) — Creating Change is a past-focused, integrated, cognitive-behavioral therapy for PTSD/SUD. It has 17 topics, which in this study were delivered in weekly one-hour sessions, in individual format. The treatment explores how PTSD and SUD arose and interacted across the patient's life, including constructing a narrative of its meaning, processing associated emotions and memories, and exploring themes related to these.
  Arms: Creating Change (CC)
Behavioral: Seeking Safety (SS) — Seeking Safety is a present-focused, evidence-based cognitive-behavioral therapy for integrated treatment of patients with PTSD/SUD. It is a cognitive-behavioral therapy comprising 25 topics, each a coping skill relevant to both disorders. In this study 17 of the 25 topics were conducted, one per weekly, one-hour, individual session.
  Arms: Seeking Safety (SS)

SUMMARY:
This study compares Creating Change, a new past-focused behavioral therapy for posttraumatic stress disorder (PTSD)/substance use disorder (SUD), to Seeking Safety, an evidence-based present-focused behavioral therapy for PTSD/SUD.

DETAILED DESCRIPTION:
This study evaluates a new behavioral therapy model, Creating Change (CC) for PTSD/SUD. CC helps clients explore the past as a step in their recovery process. It has major public health relevance in that it is a low-cost, flexible model designed for all trauma and substance abuse types, both genders, and all clinical settings. It has particular relevance for VA in that many veterans suffer from PTSD and SUD. The new model demonstrated positive results in two pilot studies.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual (DSM-IV) criteria for current PTSD and current substance use disorder
* Have used a substance in the 60 days prior to intake
* Outpatient
* Plan to stay in Boston for the next 6 months
* If on psychiatric medication, are on a stable regimen for at least 4 weeks prior to participation in the study
* Have a stable mailing address and live nearby enough to come to VA Boston for treatment
* Able to sign informed consent
* Willing to participate in all assessments and urine testing
* Willing to provide a release of information for study staff to contact treaters as needed for clinical concerns

Exclusion Criteria:

* Any current acute medical condition that would either interfere with the patient's ability to attend treatment, or would be of such severity as to affect the patient's psychological functioning
* Current bipolar I disorder, schizophrenia or other psychotic disorders, mental retardation, or organic mental disorder
* Any obvious clinical sign that the patient is not sufficiently stable to participate in the treatment, or notification by the patient's primary providers that participation would be contraindicated
* Dangerousness that would present a threat to staff or patients (e.g., history of assault within the past 6 months)
* The patient is mandated to treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Checklist total score - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  PTSD symptoms assessed via self-report measure
Change in diagnosis of PTSD on the MINI Neuropsychiatric Interview - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  PTSD diagnosis as assessed by a trained interviewer
Change in Addiction Severity Index alcohol composite score - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Alcohol use and associated problems as measured by blinded-interviewer measure Composite. These outcome variables will be measured at baseline, end of treatment and 3-month followup.
Change in Addiction Severity Index drug composite score - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Drug use and associated problems as measured by blinded-interviewer measure Composite. These outcome variables will be measured at baseline, end of treatment and 3-month followup. Urinanlysis/breathalyzer will be obtained to verify ASI self-report.

SECONDARY OUTCOMES:
Change in Quality of Life Satisfaction & Enjoyment Scale - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Self-report measure
Change in Brief Symptom Inventory-Global Severity Index - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Self-report measure
Change in Beliefs About Substance Use - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Self-report measure
Change in General Self-Efficacy - from baseline through end of treatment and 3-month followup: Self-report measure | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Self-report measure
Change in Coping Self-Efficacy Scale - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Self-report measure
Change in World Assumptions Scale - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Self-report measure
Change in Trauma Related Guilt Inventory - from baseline through end of treatment and 3-month followup | Baseline, end of treatment (approximately 4 months from baseline), and 3-month followup
  Self-report measure

CONTACTS AND LOCATIONS:
Overall Officials: Karen E. Krinsley, Ph.D., Principal Investigator — VA Boston Healthcare System; Lisa M Najavits, PhD, Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Najavits LM, Krinsley K, Waring ME, Gallagher MW, Skidmore C. A Randomized Controlled Trial for Veterans with PTSD and Substance Use Disorder: Creating Change versus Seeking Safety. Subst Use Misuse. 2018 Sep 19;53(11):1788-1800. doi: 10.1080/10826084.2018.1432653. Epub 2018 Feb 20. PMID 29461920